CLINICAL TRIAL: NCT05567159
Title: A Phase 1, Open-Label Study to Characterize the Pharmacokinetics of Donanemab Following Intravenous Doses in Healthy Participants
Brief Title: A Study of Donanemab (LY3002813) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18616; I5T-MC-AACP (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-07-01

CONDITIONS: Healthy
MeSH Terms: interventions — donanemab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Donanemab (Experimental): Participants received a 350 milligrams (mg) intravenous (IV) infusion of donanemab every two weeks for six treatment periods (1 to 6), each lasting two weeks. Treatments were administered on the first day of each period, i.e., days 1, 15, 29, 43, 57, and 71.
  Interventions: Drug: Donanemab

INTERVENTIONS:
Drug: Donanemab — Administered IV.
  Other Names: LY3002813

SUMMARY:
The main purpose of this study is to assess how fast donanemab (LY3002813) gets into the blood stream and how long it takes the body to remove it when administered as single dose in healthy participants. The study will also evaluate the safety and tolerability of donanemab. The study will last up to approximately 22 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation
* Have a body mass index (BMI) of 19.0 and 32.0, kilograms per meter squared (kg/m²), inclusive.
* Females of childbearing potential will be excluded from the study.

Exclusion Criteria:

* Have allergies to either humanized monoclonal antibodies, diphenhydramine, epinephrine, or methylprednisolone
* Have a history within the past 5 years of a primary or recurrent malignant disease
* Have used over-the-counter or prescription medications, including herbal medication, within 7 days prior to dosing
* Are pregnant or intend to become pregnant or to breastfeed during the study
* Smoke more than 10 cigarettes per day or are unable to abide by investigative site smoking restrictions
* Have a history of intracranial hemorrhage, cerebrovascular aneurysm or arteriovenous malformation, carotid, carotid artery occlusion, stroke or epilepsy or family history of dementia or Down's syndrome

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- ICON Early Phase Services Lenexa Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Donanemab
Started | 42
Received at Least One IV Infusion of Donanemab | 42
Completed | 34
Not Completed | 8
Not completed — Adverse Event | 4
Not completed — Physician Decision | 3
Not completed — Protocol deviation | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Donanemab: Participants received a 350 mg IV infusion of donanemab every two weeks for six treatment periods (1 to 6), each lasting two weeks. Treatments were administered on the first day of each period, i.e., days 1, 15, 29, 43, 57, and 71.
Arm/Group | Donanemab
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 28
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Four Weeks (AUC[0-4 Weeks]) of Donanemab (i.e) Period 2, Period 4, Period 6.
Description: As per the prespecified analysis, AUC[0-4 weeks] will be calculated as the sum of AUC0-2weeks for:
  * treatment period 1 and 2 (dosing days 1, 15 respectively) represented as period 2
  * treatment period 3 and 4 (dosing days 29, 43 respectively) represented as period 4
  * treatment period 5 and 6 (dosing days 57, 71 respectively) represented as period 6.
Time Frame: Predose, end of infusion, 24, 48, 72, 96, 168, 336 hours post-dose on days 1, 15, 29, 43, 57, 71
Population: All enrolled participants who received at least one IV infusion of donanemab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (μg*h/mL)
Arm/Group | Donanemab
Number analyzed (Participants) | 27
microgram*hour per milliliter (μg*h/mL)
  Period 2 | 17300 (23)
  Period 4 | 15400 (32)
  Period 6 | 15500 (45)

2. Primary Outcome: PK: Maximum Observed Concentration During a Dosing Interval at Steady State (Cmax, ss) of Donanemab
Description: PK: Cmax, ss of Donanemab
Time Frame: Predose, end of infusion, 24, 48, 72, 96, 168, 336 hours post-dose on day 71
Population: All enrolled participants who received at least one IV infusion of donanemab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Donanemab
Number analyzed (Participants) | 27
μg/mL | 112 (21)

3. Primary Outcome: PK: Area Under the Concentration Versus Time Curve During a Dosing Interval at Steady State (AUCτ,ss) of Donanemab
Description: PK: AUCτ,ss of Donanemab
Time Frame: Predose, end of infusion, 24, 48, 72, 96, 168, 336 hours post-dose on day 71
Population: All enrolled participants who received at least one IV infusion of donanemab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Donanemab
Number analyzed (Participants) | 27
μg*h/mL | 7590 (50)

ADVERSE EVENTS:
Time Frame: Baseline to Week 22
Description: All enrolled participants who received at least one IV infusion of donanemab.
Arm/Group | Donanemab
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 22/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donanemab (N=42)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Infusion related reaction (Injury, poisoning and procedural complications) | 7 (12)
Blood creatine phosphokinase increased (Investigations) | 3 (3)
Headache (Nervous system disorders) | 13 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT05567159/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT05567159/SAP_001.pdf